CLINICAL TRIAL: NCT05568810
Title: The Study of Adenoma Characteristics of the COX-2 and DNMT Expressions in the Index Colonoscopy to Predict the Polyp Recurrence During Surveillance
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-102-436
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Colon Polyp
Keywords: DNA methyltransferases (DNMT); cyclooxygenase-2 (COX-2)
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — polyps will be resected for IHC (immunohistochemistry) stain
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The colorectal cancer is the first incidence and ranks the third cancer-death cause in Taiwan. Based on the Taiwan-national colon cancer screening program, early colorectal cancer detection rate and the survival are markedly improved. Besides to disclose the early cancer, there are vast populations to be disclosed with colon adenoma. Some of colon adenoma really presents as advanced colon adenoma (ACA) to carry higher risk of recurrence and even cancer progression. The current clinical guidelines raise strategy for colonoscopy surveillance based on the results of the index colonoscopy to categorize the patients into different risks of colon polyp recurrence and early detection of colorectal cancer. It is worthy to validate whether the real scenario of Taiwan colonoscopy surveillance can fulfill the guidelines worldwide. Furthermore, it shall be of clinical importance to elucidate out the high risky group who may be commonly disclosed during intense colonoscopy surveillance and to disclose with advanced adenoma. Accordingly, the domestic amending to the worldwide guideline shall be in need and need a more reliable biomarker to predict the recurrence of colon adenoma during surveillance colonoscopy. Concerning, cyclooxygenase-2 (COX-2) and DNA methyltransferases (DNMT) are involved during colorectal carcinogenesis via chronic inflammatory process and early tumorigenesis. This study proposes COX-2 and DNMT shall be potential biomarkers correlating to the recurrence of colon adenoma disclosed during surveillance colonoscopy in Taiwan. We thus conduct a prospective study, containing at least 1,400 cases, who will undergo surveillance colonoscopy in National Cheng Kung University Hospital in the next year. The study shall be a large-case study to answer whether the surveillance interval of the surveillance colonoscopy can be fulfilled to the suggestion of the 2012 United States Multi-society Task Force (USMTF) on colorectal cancer guideline. Factors that affect the detection of polyps in the surveillance will be explored. Based on the invitation of the patients to receive surveillance colonoscopy, the study also test whether COX-2 or DNMT over-expression are markers to predict polyps recurrence and to identify the risky patient deserve for earlier colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive surveillance colonoscopy during the study period at National Cheng Kung University Hospital, a tertiary referral medical center in Taiwan, are enrolled in the study

Exclusion Criteria:

* poor bowel preparation, failed cecal intubation, contraindication for biopsy or polypectomy, patients with a history of inflammatory bowel disease, and those who are under 18 years old, decline to join the study, or do not have previous colonoscopy conducted in our institute

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who receive surveillance colonoscopy during the study period at National Cheng Kung University Hospital, a tertiary referral medical center in Taiwan, are enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
the compatibility of surveillance colonoscopy with the USMTF guideline in Taiwan | usual the exam of colonoscopy: 10 min to 60 min
  To determine the compatibility of surveillance colonoscopy with the USMTF guideline for different histological features of colon adenoma at index colonoscopy in Taiwan
Factors that affect the detection of polyps in the surveillance | usual the exam of colonoscopy: 10 min to 60 min
  To explore factors that affect the detection of polyps in the surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Ying Chen, MD, Principal Investigator — National Cheng-Kung University Hospital